CLINICAL TRIAL: NCT00487162
Title: The Association Between Peri-Operative Hyperglycemia and Major Morbidity and Mortality
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: potential harm of insulin infusion outweights the benefit.
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120070093
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-09

CONDITIONS: Hyperglycemia
Keywords: glycemic control, diabetes, obesity, comorbidities
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensive glycemic control (Experimental): In the intensive treatment group, continuous insulin infusion (50 IU of Novolin R [Novo Nordisk]) in 50ml of 0.9% saline via infusion pump will be started when the blood glucose level exceeds 110 mg / dL on two consecutive samples and will be adjusted to maintain the blood glucose level between 80 and 110 mg / dL. If the glucose level falls below 80 mg / dL, the insulin infusion will be tapered and discontinued.
  Interventions: Procedure: intensive glycemic control
- conventional glycemic control (Active Comparator): In this group if the subject's blood glucose level should exceed 200 mg/dL the subject will be treated with a continuous insulin infusion to maintain blood glucose levels between 180-200mg/dL
  Interventions: Drug: conventional glycemic control

INTERVENTIONS:
Procedure: intensive glycemic control — intravenous insulin titrated every 30 minutes to serum glycemic level of 80-100mg/dl
  Other Names: Novo Regular Insulin
  Arms: intensive glycemic control
Drug: conventional glycemic control — Novo regular insulin administered when glucose level exceeded 200 mg/dl and titrated to maintain level between 180-200 mg/dl
  Arms: conventional glycemic control

SUMMARY:
Surgery induces a stress effect on the body partially through a catabolic energy state. In turn, glucose levels may rise to levels which have been associated with major morbidity (Golden, 1999) and mortality (Ouattara, 2005). An increasing body of evidence suggests that intensive insulin therapy for tight control of blood glucose levels in certain surgical and critical care patient populations may improve mortality and selected morbidity outcomes when compared to those patients receiving conventional insulin therapy and blood glucose management. More specifically, poor intra-operative blood glucose control is associated with worse outcome after cardiac surgery. Intensive insulin therapy with tight blood glucose control in surgical patients while in the ICU may reduce morbidity and mortality. Such outcome improvements would clearly provide benefits to patients, providers and payers. To date, there is scant research examining whether intensive insulin therapy for tight control of blood glucose in the perioperative period can alter outcomes for the non cardiac surgery population. The purpose of this study is to determine whether intensive insulin therapy for tight control of blood glucose in the perioperative period in non cardiac major surgery patients is associated with altered morbidity and mortality rates.

DETAILED DESCRIPTION:
Intensive insulin therapy to control blood glucose levels reduces morbidity and mortality in intensive care unit patients and in cardiac surgical patients but its role in patients undergoing non-emergent non-cardiac surgery is unknown. Benefits of glucose control may result from prevention of immune system dysfunction, reduction in systemic inflammation, and protection of endothelium and mitochondrial structure and function, all of which are known to be altered by high stress states such as that induced by surgical procedures.

In a prospective, randomized, controlled study of adult patients admitted to our operating suite for non-emergent non-cardiac surgery, we propose to correlate in-hospital morbidity and mortality with blood glucose levels of patients who are expected to have moderate to high levels of physiologic stress as a result of their pre-existing medical conditions or as a result of the proposed surgical procedure. Specifically, patients who are deemed to be American Society of Anesthesiologists Risk Classification 1-3 or higher, or patients undergoing intermediate and high risk procedures shall be considered to have moderate to high physiologic stress.

Determination of intermediate / high risk procedures shall be according to the American College of Cardiology / American Heart Association 2002 Guidelines for Perioperative Cardiovascular Evaluation for Noncardiac Surgery as outlined in Table 1.

Table 1. Cardiac Event Risk Stratification for Noncardiac Surgical Procedures High (Reported cardiac risk often >5%)

* Emergent major operations, particularly in the elderly
* Aortic and other major vascular surgery
* Peripheral vascular surgery
* Anticipated prolonged surgical procedures associated with large fluid shifts and/or blood loss Combined incidence of cardiac death and nonfatal myocardial infarction. Further preoperative cardiac testing is not generally required. Intermediate (Reported cardiac risk generally <5%)
* Intraperitoneal and intrathoracic surgery
* Carotid endarterectomy surgery
* Head and neck surgery
* Orthopedic surgery
* Prostate surgery Low (Reported cardiac risk generally <1%):
* Endoscopic procedures
* Superficial procedures
* Cataract surgery
* Breast surgery

Prior to entering the operating suite for surgery, patients will be randomly assigned to receive either intensive insulin treatment or conventional insulin treatment. Treatment assignment will be performed using sealed envelopes, and patients stratified according to Table 2.

TABLE 2. Baseline Characteristics of Patients. Variable Intention to Treat Group P Value Male sex (%) Age (Years) Type of Surgery

* Intracranial (%)
* Head & Neck (%)
* Thoracic (%)
* Vascular (%)
* Gastrointestinal (%)
* Urologic (%)
* Orthopedic (%)
* Gynecologic (%)
* Myocutaneous (%) History of Cancer (%) History of Organ Failure before Surgery (%) Organ Failure After Surgery (%) History of Diabetes (%)
* Treated with insulin
* Treated with oral diabetic agent, diet or both

Inclusion criteria:

* Patients scheduled for non emergent surgery under either general or regional anesthesia deemed to have moderate to high physiologic stress
* Male and female subjects over the age of 18 with or without a diagnosis of diabetes mellitus
* Patients must be able to provide informed consent

Exclusion criteria:

* Cognitively impaired
* Non-English or Spanish speaking with no relative present who is fluent in reading and comprehending English or Spanish.
* Female patients of child bearing age who have a positive pregnancy test on admission.

In all patients, whole blood hemoglobin A1C and glucose levels will be drawn prior to induction of anesthesia. Additional whole blood glucose levels will be drawn at the time of induction of anesthesia, at skin incision, hourly throughout the operation, at emergence from anesthesia, every hour up to three hours after the completion of surgery, and then once per day until the patient is discharged from the hospital.

In the intensive treatment group, continuous insulin infusion (50 IU of Novolin R [Novo Nordisk]) in 50mL of 0.9% saline via infusion pump will be started when the blood glucose level exceeds 110 mg/dL and will be adjusted to maintain the blood glucose level between 80 and 110 mg/dL. Adjustments will be made according to the University Hospital's ICU Adult Insulin Infusion Protocol. When the blood glucose level falls below 80 mg/dL, the insulin infusion will be tapered and discontinued. For patients going to the ICU after surgery, insulin infusions will be continued according to the University Hospital's ICU Adult Insulin Infusion Protocol under the direction of the ICU staff. For patients not being to the ICU after surgery, insulin infusions will be tapered to off after the final hourly blood glucose determination at three hours after the completion of surgery. The University Hospital's Blood Glucose Management Order Set for Medical and Surgical Patients will then be adopted for continued glucose management.

In the conventional treatment group, continuous insulin infusion will be started when the blood glucose level exceeds 200 mg/dL and will be adjusted to maintain the blood glucose level between 180 and 200 mg/dL. Adjustments will be made according to a modified ICU Adult Insulin Infusion Protocol. When the blood glucose level falls below 180mg/dL, the insulin infusion will be tapered and discontinued. For patients transferred to an ICU after surgery, insulin infusions will be continued according to the University Hospital's ICU Adult Insulin Infusion Protocol under the direction of the ICU staff. For patients not being transferred to an ICU after surgery, insulin infusions will be tapered to off after the final hourly blood glucose determination at three hours after the completion of surgery. The University Hospital's Blood Glucose Management Order Set for Medical and Surgical Patients will then be adopted for continued glucose management.

How will the study be analyzed?

At baseline, data on demographic and clinical characteristics of the patients (see Table 1) will be obtained. Blood will be systematically sampled and whole blood glucose levels determined as described above. All blood glucose values will be tabulated from baseline through end of study.

A research associate blinded to the treatment groups will determine morbidity and mortality by reviewing the patient's medical record upon discharge from the hospital and recording the occurrence of morbidity and mortality by the following criteria:

1. Post-operative surgical wound infection - a clinical condition requiring antibiotic treatment beyond the UH Surgical Infection Prevention (SIP) protocol and / or subsequent wound drainage / debridement
2. Systemic infection - presence of bacteremia or prolonged (i.e. greater than 10 days) use of antibiotics
3. Myocardial Injury - postoperative EKG changes that reveal new Q waves or S-T segment elevations greater than 1mm in any lead(s) or serum troponin levels that exceed….
4. Malignant arrhythmia - asystole, ventricular tachycardia or fibrillation requiring cardiopulmonary resuscitation, antiarrhythmia therapy, or defibrillator implantation
5. Respiratory Injury - mechanical ventilation for more than 48 hours, reintubation, or planned tracheostomy
6. Neurological Injury - focal brain injury with permanent functional deficit, irreversible encephalopathy
7. Renal Injury - a level of serum creatinine twice that present on admission to the hospital or acute renal failure requiring dialysis
8. Hepatic Injury - bilirubin level of >3mg per deciliter
9. Venous Thromboembolism - deposition of thrombus in peripheral or central veins as determined by Doppler ultrasonography, angiography or computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for non emergent surgery under either general or regional anesthesia deemed to have moderate to high physiologic stress
* Male and female subjects over the age of 18 with or without a diagnosis of diabetes mellitus
* Patients must be able to provide informed consent

Exclusion Criteria:

* Cognitively impaired
* Non-English or Spanish speaking with no relative present who is fluent in reading and comprehending English or Spanish.
* Female patients of child bearing age who have a positive pregnancy test on admission.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Jeffery Freda, MD, MBA, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Furnary AP, Gao G, Grunkemeier GL, Wu Y, Zerr KJ, Bookin SO, Floten HS, Starr A. Continuous insulin infusion reduces mortality in patients with diabetes undergoing coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2003 May;125(5):1007-21. doi: 10.1067/mtc.2003.181. PMID 12771873
- [Background] Ouattara A, Lecomte P, Le Manach Y, Landi M, Jacqueminet S, Platonov I, Bonnet N, Riou B, Coriat P. Poor intraoperative blood glucose control is associated with a worsened hospital outcome after cardiac surgery in diabetic patients. Anesthesiology. 2005 Oct;103(4):687-94. doi: 10.1097/00000542-200510000-00006. PMID 16192760

RESULTS

PARTICIPANT FLOW:
Recruitment Details: enrollment period 6/07-3/09. potential subjects were recruited from the pre-operative admission unit and were screened if there ages were 18-90,undergoing general anesthesia for surgical procedures greater than 2 hours.
Pre-assignment Details: Subjects were randomized to a specific study arm based on a computer generated randomization table. 49 participants are included in the baseline characteristic module because although 56 signed consent, some subjects withdrew the consent prior to study procedures and several withdrawn by attending anesthesiologist.
Groups:
- Conventional Glycemic Control: Subjects randomized to this study arm had their glucose levels monitored hourly and if the result was greater than 200mg/dL their anesthesia care provider was notified. The subject was treated as to thie care provider discretion.
- Intensive Glycemic Control: In the intensive treatment group, continuous insulin infusion (50 IU of Novolin R [Novo Nordisk]) in 50ml of 0.9% saline via infusion pump will be started when the blood glucose level exceeds 110 mg / dL on two consecutive samples and will be adjusted to maintain the blood glucose level between 80 and 110 mg / dL. Adjustments will be made according to the University Hospital's ICU Adult Insulin Infusion Protocol - modified 10/1/07 (Appendix A). When the blood glucose level falls below 80 mg / dL, the insulin infusion will be tapered and discontinued. For patients going to the ICU after surgery, insulin infusions will be continued according to the University Hospital's ICU Adult Insulin Infusion Protocol under the direction of the ICU staff. For patients not being to the ICU after surgery, insulin infusions will be tapered to off after the final hourly blood glucose determination at three hours after the completion of surgery.
Period: Overall Study
Arm/Group | Conventional Glycemic Control | Intensive Glycemic Control
Started | 30 | 26
Completed | 28 | 21
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: males and females between the ages of 18 and 89.
Groups:
- Conventional Glycemic Control: Subjects randomized to this study arm had their glucose levels monitored hourly and if the result was greater than 200 mg/dL their anesthesia care provider was notified. The subject was treated as to their care provider discretion.
- Intensive Glycemic Control: In this treatment group, continuous insulin infusion (50 IU of Novolin R [Novo Nordisk]) in 50mL of 0.9% saline via infusion pump will be started when the blood glucose level exceeds 110 mg/dL and will be adjusted to maintain the blood glucose level between 80 and 110 mg/dL.
- Total: Total of all reporting groups
Arm/Group | Conventional Glycemic Control | Intensive Glycemic Control | Total
Number analyzed (Participants) | 28 | 21 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 20 | 45
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Wound Infection
Time Frame: 7-10 days post op
Population: no analysis was done as the study was terminated due to patient safety concerns
Groups:
- Strict Glycemic Control: strict glycemic control: intravenous insulin titrated every 30 minutes to serum glycemic level of 80-100mg/dl
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hemodynamic Instability
Time Frame: 0-48 hours post op
Population: no analysis was done as the study was terminated due to patient safety concerns
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Conventional Glycemic Control: Subjects randomized to this study arm had their glucose levels monitored hourly and if the result was greater than 200mg/dL their anesthesia care provider was notified. The subject was treated as to their care provider discretion.
- Intensive Glycemic Control: Subjects randomized to this group had glucose levels monitored hourly and when >110mg/dL an insulin drip was initiated to maintain glucose levels between 80-110
Arm/Group | Conventional Glycemic Control | Intensive Glycemic Control
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/21
Other Adverse Events (participants affected / at risk) | 0/28 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Glycemic Control (N=28) | Intensive Glycemic Control (N=21)
hypoglycemia (Endocrine disorders) | 0 | 1 — subject's serum blood glucose level dropped to <60. Insulin discontinued

LIMITATIONS AND CAVEATS:
Study was terminated. No final conclusion drawn. A sentinel article was published in Feb 2009 issue of Anesthesiology which questioned the safety of intense insulin therapy/strict glycemic control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No